CLINICAL TRIAL: NCT01807598
Title: A Study of Brentuximab Vedotin (SGN-35) in CD30-Positive Systemic Mastocytosis With or Without an Associated Hematological Clonal Non-Mast Cell Lineage Disease (AHNMD)
Brief Title: Brentuximab Vedotin in Treating Patients With Advanced Systemic Mastocytosis or Mast Cell Leukemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Jason Robert Gotlib (Other)
Collaborators: Seagen Inc. (Industry)
Responsible Party: Sponsor-Investigator, Jason Robert Gotlib, Professor of Medicine (Hematology), Stanford University
Organization: Stanford University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-25727; NCI-2013-00537 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); IRB-25727 (Other: Stanford IRB); 107011 (Other Grant/Funding Number: Seattle Genetics); HEMMPD0016 (Other: OnCore)
Record Dates: First submitted 2013-03-05; First posted 2013-03-08 (Estimated); Results first posted 2019-01-29 (Actual); Last update posted 2019-01-29 (Actual); Status verified 2019-01

CONDITIONS: Aggressive Systemic Mastocytosis; Mast Cell Leukemia; Systemic Mastocytosis
MeSH Terms: conditions — Mastocytosis, Systemic; Leukemia, Mast-Cell | interventions — Brentuximab Vedotin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Brentuximab vedotin (Experimental): Subjects receive a 30-minute IV infusion of brentuximab vedotin once every 21 days for 8 courses, in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Brentuximab vedotin

INTERVENTIONS:
Drug: Brentuximab vedotin
  Other Names: Adcetris; anti-CD30 antibody-drug conjugate; anti-CD30 ADC; SGN-35

SUMMARY:
This pilot clinical trial studies brentuximab vedotin in treating patients with advanced systemic mastocytosis or mast cell leukemia. Monoclonal antibodies, such as brentuximab vedotin, can block cancer growth in different ways. Some block the ability of cancer cells to grow and spread. Others find cancer cells and help kill them or carry cancer-killing substances to them

DETAILED DESCRIPTION:
Brentuximab vedotin is an antibody with a covalently attached toxin. The antibody portion targets the protein CD30 on the surface of cells, and the toxin acts against those cells.

PRIMARY OBJECTIVES:

I. To evaluate the response rate to SGN-35 (brentuximab vedotin) in patients with tumor necrosis factor receptor superfamily, member 8 (CD30+) advanced systemic mastocytosis (SM) (ASM or mast cell leukemia [MCL] with or without an associated hematological clonal non-mast cell lineage disease [AHNMD]).

SECONDARY OBJECTIVES:

I. To evaluate the tolerability and safety profile of SGN-35 in patients with SM.

II. To evaluate expression of CD30 on neoplastic mast cells before and during therapy with SGN-35.

III. To evaluate changes in mastocytosis related symptom scores and quality of life (QOL) using a modified Myeloproliferative Neoplasm Symptom Assessment Form (MPNSAF).

IV. To evaluate the duration of response (DoR) and time to response (TTR). V. To evaluate progression-free survival (PFS).

OUTLINE:

Patients receive brentuximab vedotin intravenously (IV) over 30 minutes on day 1. Treatment repeats every 21 days for 8 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 6 weeks for 1 year and then every 12 weeks thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-3
* Life expectancy > 12 weeks
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) =< 2.5 x upper limit of normal (ULN), if caused by ASM/MCL =< 5 x ULN
* Serum direct bilirubin =< 1.5 x ULN; if considered related to ASM/MCL =< 3 x ULN
* Serum creatinine =< 2.0 mg/dL
* A diagnosis of systemic mastocytosis (SM) per 2008 World Health Organization (WHO) Criteria
* Neoplastic mast cells must express CD30 by immunohistochemistry or flow cytometry
* At least one of the eligible organ damage findings as defined by the international consensus response criteria
* Females of childbearing potential and males who have partners of childbearing potential must agree to use an effective contraceptive method during the study and for 30 days following the last dose of study drug
* Females of childbearing potential must have a negative serum or urine beta-human chorionic gonadotropin (hCG) pregnancy test result within 7 days prior to the first dose of SGN-35
* Females of non-childbearing potential are those who are postmenopausal greater than 1 year or who have had a bilateral tubal ligation or hysterectomy

Exclusion Criteria:

* Unwilling or unable to comply with the protocol
* Any other concurrent severe known disease (except carcinoma in-situ) or concurrent severe and/or uncontrolled medical condition (e.g. uncontrolled diabetes, or active uncontrolled infection) which could compromise participation in the study
* History of another primary malignancy that has not been in remission for at least 3 years (the following are exempt from the 3-year limit: non-melanoma skin cancer, fully excised melanoma in situ [stage 0], curatively treated localized prostate cancer, and cervical carcinoma in situ on biopsy or a squamous intraepithelial lesion on Papanicolaou [PAP] smear)
* Cardiovascular disease including congestive heart failure grade III or IV according to the New York Heart Association (NYHA) classification, left ventricular ejection fraction of < 50%, myocardial infarction within previous 6 months or poorly controlled hypertension
* Pregnant or lactating
* Neuropathy greater than or equal to grade 2
* Known hypersensitivity to any excipient contained in the drug formulation
* Confirmed diagnosis of human immunodeficiency virus (HIV) infection or active viral hepatitis
* Presenting with an AHNMD requiring immediate cytoreductive therapy or targeted drugs (eg, AML)
* Received any investigational agent, chemotherapy, interferon-alfa, or 2-chlorodeoxyadenosine (2-CdA, cladribine) within 30 days prior to Day 1
* Received hematopoietic growth factor support within 14 days of Day 1 of SGN-35
* Use of prednisone (or equivalent corticosteroid dose) for SM up to 10 mg/day or its equivalent is allowed, but it cannot have been started during screening; patients who are on prednisone up to 10 mg/day for medical problems unrelated to SM are also permitted on study
* Presence of FIP1L1-PDGFR-alpha fusion even with resistance to imatinib
* Received any treatment with SGN-35 prior to study entry
* Any surgical procedure within 14 days of Day 1, excluding central venous catheter placement or other minor procedures (eg, skin biopsy)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2013-09; Primary Completion 2017-09 (Actual); Study Completion 2017-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jason Gotlib, Principal Investigator — Stanford University Hospitals and Clinics
Locations (2):
- United States (2):
  - Stanford University, School of Medicine, Stanford, California
  - MD Anderson Cancer Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gotlib J, Baird JH, George TI, Langford C, Reyes I, Abuel J, Perkins C, Schroeder K, Bose P, Verstovsek S. A phase 2 study of brentuximab vedotin in patients with CD30-positive advanced systemic mastocytosis. Blood Adv. 2019 Aug 13;3(15):2264-2271. doi: 10.1182/bloodadvances.2019000152. PMID 31350306

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Brentuximab Vedotin
Started | 10
Completed | 4
Not Completed | 6
Not completed — Withdrawal by Subject | 4
Not completed — Adverse Event | 1
Not completed — Other Physician Decision | 1

BASELINE CHARACTERISTICS:
Arm/Group | Brentuximab Vedotin
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 4
  >=65 years | 6
Age, Continuous [Mean (Full Range); unit: Years] | 65.8 [37.8 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 10
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 9
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 10

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate (ORR) Per Consensus International Response Criteria (Rate of Complete or Partial Remissions or Clinical Improvement)
Description: Overall response rate (ORR) is sum of complete response (CR); partial response (PR); and clinical improvement (CI) in 1 year, ie, ORR=CR+PR+CI. The outcome is the number of participants without dispersion.
  CR is following with response duration(RD) ≥12 weeks (wk)
  * No mast cell disease
  * Tryptase <20 ng/mL
  * Neutrophils ≥1x10e9/L with normal differential
  * Hemoglobin ≥11 g/dL
  * Platelets ≥100x10e9/L
  * No hepatosplenomegaly
  * No systemic mastocytosis(SM)-related organ damage PR is following with RD ≥12wk
  * Neither CR or progressive disease(PD)
  * Neoplastic mast cells reduced ≥50%
  * Tryptase reduced ≥50%
  * 1+ disease finding resolved CI is following with RD ≥12wk
  * Neither CR; PR; or PD
  * 1+ of findings above Stable disease (SD) Not CR, PR, Cl, or PD Progressive disease (PD)
  Any of:
  * Worsening organ damage
  * Doubling of laboratory abnormality
  * New transfusion dependence of ≥4 units red cells or platelets at 8wk
    •+ ≥100% in transfusions for 8wk
  * 10-cm+ splenomegaly
Time Frame: Up to 1 year
Population: 1 of 10 participants were not evaluable due to early death during Cycle 1 (considered unrelated to study treatment)
Measure: Number; unit: participants
Arm/Group | Brentuximab Vedotin
Number analyzed (Participants) | 9
participants | 0

2. Secondary Outcome: Brentuximab Vedotin Toxicity
Description: Toxicity was assessed as the number of adverse events considered possibly, probably, or definitely-related to treatment with brentuximab vedotin. The outcome is reported as the total number of related events, a number without dispersion, and the number of related events (without dispersion) considered to be either a hematologic toxicity or non-hematologic toxicity.
Time Frame: Up to 1 year
Measure: Number; unit: Related adverse events
Arm/Group | Brentuximab Vedotin
Number analyzed (Participants) | 10
Related adverse events
  Total related adverse events (toxicities) | 36
  Related hematologic toxicity | 12
  Related non-hematologic toxicity | 24

3. Secondary Outcome: Percent Change of CD30 Expression on Neoplastic Mast Cells
Description: The presence of the CD30 marker (epitope) on neoplastic (cancerous) mast cells in core bone marrow biopsy samples was assessed by immunohistochemical methods, before and after brentuximab vedotin treatment. CD30 is a member of the TNF-receptor (TNF-R) superfamily, and is a transmembrane glycoprotein receptor that is normally at very low levels on the surface of activated T-cells. Overexpression of the CD30 marker is indicative of T-cell lymphoproliferative disorders and neoplastic mast cells, and the effect of a particular treatment on CD30 expression may be related to the efficacy of that treatment. The outcome is reported as the median percentage change in the level of CD30 detected, reported with full range.
Time Frame: Baseline and up to 1 year
Population: CD30 marker data was not obtained for some participants.
Measure: Median (Full Range); unit: percentage change in CD30+ cells
Arm/Group | Brentuximab Vedotin
Number analyzed (Participants) | 8
percentage change in CD30+ cells | -1 [-62 to 45]

4. Secondary Outcome: Myeloproliferative Neoplasm Symptom Assessment Form (MPN-SAF) Total Symptom Score
Description: The clinical effect of patient symptoms associated with systemic mastocytosis or mast cell leukemia were assessed with the patient-reported outcome survey entitled Myeloproliferative Neoplasm Symptom Assessment Form with Mast Cell Disorder Symptoms [(MPN-SAF(MCD)]. The MPN-SAF(MCD) is a 36-question survey, with possible responses ranged from 0 to 10, with 0 indicating not present or no effect; 1 meaning present but most favorable; and 10 meaning worst imaginable (least favorable). Total range is 0 to 360, with 0 being best possible, and 360 being worst possible. Total symptom score is calculated as the sum of the individual survey scores reported at baseline and after treatment, with lower numbers indicating less effect, and larger numbers indicated greater effect. The outcome is reported as mean score value with dispersion.
Time Frame: Up to 1 year
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Brentuximab Vedotin
Number analyzed (Participants) | 10
score on a scale
  Baseline (Pre-treatment) | 36.2 (18.1)
  After Treatment | 23.6 (15.6)

5. Secondary Outcome: Quality of Life (QoL) Score Using a Modified Myeloproliferative Neoplasm Symptom Assessment Form (MPN-SAF)
Description: Overall quality of life (QoL) was assessed by a single specific question from the 36-question Myeloproliferative Neoplasm Symptom Assessment Form with Mast Cell Disorder Symptoms [(MPN-SAF(MCD)] survey. Possible responses for theQoL question range from 0 to 10, with 0 indicating "as good as it can be" (most favorable), and 10 meaning "as bad as it can be" (least favorable). The QoL score was obtained at baseline and after treatment. The outcome is reported as mean score with dispersion.
Time Frame: Up to 1 year
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Brentuximab Vedotin
Number analyzed (Participants) | 10
score on a scale
  Baseline (Pre-treatment) | 5 (2.7)
  After Treatment | 2.6 (2.7)

6. Secondary Outcome: Duration of Response (DOR)
Description: Duration of response (DOR) is defined as the time from the start of the first confirmed response until the date of the first documented and confirmed disease progression or death due to ASM or MCL. For participants with a confirmed clinical response, the outcome was to be reported as the median DOR with standard deviation.
Time Frame: Up to 1 year
Population: Duration of response (DOR) can not be determined if no participants had a response.
Arm/Group | Brentuximab Vedotin
Number analyzed (Participants) | 0

7. Secondary Outcome: Time to Response (TTR)
Description: Time to response (TTR) is defined as the time from the date of start of treatment to the date of first confirmed response. For participants with a confirmed clinical response, the outcome was to be reported as the median TTR with standard deviation.
Time Frame: Up to 1 year
Population: Time to response (TTR) can not be determined if no participants had a response.
Arm/Group | Brentuximab Vedotin
Number analyzed (Participants) | 0

8. Secondary Outcome: Progression-free Survival (PFS)
Description: Progression-free survival (PFS) is defined as the time from the date of start of treatment until disease progression; death; or initiation of new therapy. The outcome is reported as the mean number of days of PFS, with 95% confidence interval.
  Progressive disease (PD) is any of the following:
  * Worsening of any organ damage
  * Doubling of any laboratory abnormality
  * New transfusion dependence of ≥ 4 units red cells or platelets at 8 wk
  * ≥ 100% increase in transfusions for 8 wk
  * 10-cm+ splenomegaly
Time Frame: Up to 1 year
Measure: Mean (95% Confidence Interval); unit: Days
Arm/Group | Brentuximab Vedotin
Number analyzed (Participants) | 10
Days | 210 [77 to 343]

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Brentuximab Vedotin
All-Cause Mortality (participants affected / at risk) | 1/10
Serious Adverse Events (participants affected / at risk) | 4/10
Other Adverse Events (participants affected / at risk) | 10/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Brentuximab Vedotin (N=10)
Intracranial hemorrhage (Nervous system disorders) | 1 (1)
Portal vein thrombosis (Hepatobiliary disorders) | 1 (1)
Respiratory, thoracic and mediastinal disorders - Other, Epiglottitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Brentuximab Vedotin (N=10)
Neutropenia (Blood and lymphatic system disorders) | 3 (11)
Anemia (Blood and lymphatic system disorders) | 2 (3)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1)
Fatigue (General disorders) | 4 (9)
Abdominal Pain (Gastrointestinal disorders) | 2 (4)
Anorexia (Metabolism and nutrition disorders) | 2 (3)
Constipation (Gastrointestinal disorders) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Depression (Psychiatric disorders) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 2 (3)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Infusion Related Reaction (General disorders) | 2 (5)
Rash (Skin and subcutaneous tissue disorders) | 2 (4)
Vomiting (Gastrointestinal disorders) | 2 (3)
Ascites (Gastrointestinal disorders) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Oral pain (Gastrointestinal disorders) | 1 (1)
Edema limbs (General disorders) | 1 (1)
Fever (General disorders) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1)
Sinusitis (Infections and infestations) | 1 (1)
Upper respiratory infection (Infections and infestations) | 1 (1)
Vaginal infection (Infections and infestations) | 1 (1)
Wound infection (Infections and infestations) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (2)
Insomnia (Psychiatric disorders) | 1 (1)
Ear pain (Ear and labyrinth disorders) | 1 (1)
Watering eyes (Eye disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Urinary frequency (Renal and urinary disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-04-03): https://cdn.clinicaltrials.gov/large-docs/98/NCT01807598/Prot_SAP_000.pdf